CLINICAL TRIAL: NCT03904329
Title: Obesity Paradox in Non Valvular Atrial Fibrillation
Brief Title: Obesity Paradox in Non Valvular Atrial Fibrillation Regarding Outcomes: Fact or Fiction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christena amir, Principal investigator, Assiut University
Other Study IDs: Assuit35
Record Dates: First submitted 2019-03-25; First posted 2019-04-05 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-02

CONDITIONS: Obesity Paradox
MeSH Terms: interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese Patients with non valvular AF: Obese Patients with non valvular AF using oral anti coagulants
  Interventions: Drug: Oral Anticoagulant

INTERVENTIONS:
Drug: Oral Anticoagulant — Oral tablets of anti coagulations either warfare or NOACs

SUMMARY:
Obesity paradox In patient with non valvular atrial fibrillation

DETAILED DESCRIPTION:
Study role of obesity in outcomes of anticoagulation in patients with non valvular atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* patients presented with non valvular AF
* patients on oral anticoagulant

Exclusion Criteria:

* valvular AF
* Mental illness
* History of cerebrovascular stroke
* history of bleeding tendency
* history of Chronic renal failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with non valvular atrial fibrillation within one year from 1/6/2019 to 31/5/2020 among patients with non valvular in assuit university hospitals
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between obesity and outcomes in non valvular atrial fibrillation | Sixth months
  To study effect of obesity in outcomes of non valvular atrial fibrillation regarding the effect of obesity in the outcome of anticoagulants

CONTACTS AND LOCATIONS:
Locations (1):
- Kristen amir, Asyut, Egypt